CLINICAL TRIAL: NCT07080307
Title: Artificial Intelligence-Based Predictive Models for Estimating Treatment Response in Sciatica Patients Treated With Transforaminal Epidural Steroid Injection (TFESI)
Brief Title: Artificial Intelligence (AI)-Based Prediction of Treatment Response in Sciatica Patients Receiving Transforaminal Epidural Steroid Injection
Status: Not yet recruiting | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: MAR.FTR.FK.01
Record Dates: First submitted 2025-07-15; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Sciatica; Low Back Pain; Lumbar Spinal Stenosis; Radiculopathy; Lumbar Disc Herniation
Keywords: sciatica, radiculopathy, lumbar disc herniation, spinal stenosis, low back pain
MeSH Terms: conditions — Sciatica; Low Back Pain; Spinal Stenosis; Radiculopathy; Intervertebral Disc Displacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This prospective observational study aims to develop artificial intelligence (AI)-based predictive models to estimate treatment response in patients with sciatica undergoing transforaminal epidural steroid injection (TFESI). Approximately 1500 adult patients diagnosed with sciatica and scheduled for TFESI at Marmara University Training and Research Hospital Algology Clinic will be enrolled. Clinical, radiological, laboratory, and psychological data will be systematically collected before the procedure and at multiple follow-up points (1 hour, 3 weeks, 3 months, and 6 months post-treatment). Pain relief, measured by a 50% or greater reduction in the Numeric Rating Scale (NRS), will be the primary outcome. The study will use these comprehensive data sets to train and validate AI algorithms, aiming to create a decision-support system that can predict individual patient responses to TFESI and improve personalized treatment planning.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Presence of clinical and radiological radiculopathy findings consistent with L4, L5, or S1 nerve root involvement
* Symptoms present for at least 3 months
* Resistant to conservative treatment
* Scheduled for transforaminal epidural steroid injection (TFESI) by a pain medicine specialist
* Being willing to participate in the study and having signed a consent form

Exclusion Criteria:

* Malignancy
* Coagulation disorders
* Pregnancy
* History of allergic reaction to the injected substances
* History of major psychiatric disorders
* Presence of known coagulopathy
* Receiving systemic steroid treatment for any reason
* Having received an epidural steroid injection within the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from the Algology Clinic of Marmara University Pendik Training and Research Hospital. The population includes patients who have been referred for transforaminal epidural steroid injection (TFESI) as part of routine clinical care for sciatica. Data will be collected prospectively during their treatment and follow-up visits.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Change in pain intensity measured by Numeric Rating Scale (NRS) | Baseline, 1 hour, 3 months, 6 months after TFESI
  Pain intensity will be assessed using the Numeric Rating Scale (0-10). A reduction of ≥50% from baseline will be considered a positive treatment response.
Change in functional status measured by Oswestry Disability Index (ODI) | Baseline, 3 months, 6 months
  Functional disability will be assessed using the validated ODI questionnaire.

SECONDARY OUTCOMES:
Change in psychological status measured by Beck Depression Inventory (BDI) | Depression symptoms will be evaluated using BDI to assess changes related to pain improvement.
  Baseline, 3months and 6 months
Change in health-related quality of life measured by SF-12 | Baseline, 3 months and 6 months
  SF-12 will be used to assess the impact of pain and treatment on quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara Üniversitesi Tıp Fakültesi, İstanbul , Maltepe 34854 Recruiting, Istanbul, Maltepe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No